CLINICAL TRIAL: NCT05257967
Title: CSF Liquid Biopsy Based Characterization of Leptomeningeal Disease in EGFR Mutant Non-Small Cell Lung Cancer
Brief Title: CSF Analysis in EGFR Mutant Non-Small Cell Lung Cancer with Leptomeningeal Disease
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: British Columbia Cancer Agency (Other)
Responsible Party: Principal Investigator, Cheryl, Prinicipal Investigator, British Columbia Cancer Agency
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: LUEGFRLM
Record Dates: First submitted 2022-02-05; First posted 2022-02-25 (Actual); Last update posted 2025-02-11 (Actual); Status verified 2025-02

CONDITIONS: EGFR Activating Mutation; Leptomeningeal Metastasis; Non Small Cell Lung Cancer
Keywords: non-small cell lung cancer; EGFR; leptomeningeal disease
MeSH Terms: conditions — Meningeal Carcinomatosis; Carcinoma, Non-Small-Cell Lung; Meningeal Neoplasms | interventions — Spinal Puncture; Phlebotomy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Experimental arm (Experimental): ddPCR and BC Cancer NGS panel completed on cerebral spinal fluid and blood circulating tumor DNA
  Interventions: Diagnostic Test: Lumbar puncture and Phlebotomy

INTERVENTIONS:
Diagnostic Test: Lumbar puncture and Phlebotomy — Sampling of cerebral spinal fluid and plasma.

SUMMARY:
Leptomeningeal disease is malignant seeding of the leptomeninges and presents with a variety of symptoms frequently impacting quality of life. With improvement in treatment options, rates of leptomeningeal disease are increasing and currently found in up to 9% of EGFR mutant NSCLC.

Systemic therapy may be more effective if it can target the correct molecular aberration. The molecular characterization of central nervous system disease may differ from disease outside of the central nervous system. The aim of this pilot trial is to evaluate for molecular differences between cerebral spinal fluid (CSF) and blood circulating tumor DNA (ctDNA) through the use of ddPCR and BC Cancer NGS panel molecular testing.

DETAILED DESCRIPTION:
The aim of this pilot trial is to evaluate the concordance/discordance of molecular profiling of CSF and plasma ctDNA after the development of leptomeningeal disease in EGFR mutant NSCLC. Patients with EGFR mutant NSCLC who develop leptomeningeal disease on a first, second or third generation tyrosine kinase inhibitor are potentially eligible for this clinical trial.

This is a prospective pilot study designed to accrue 10 patients. Baseline MRI brain and spine must be completed prior to enrolment to insure that a lumbar puncture can be completed safely. All eligible subjects will be consented for ddPCR and Canexia Follow It plasma and CSF based molecular testing. Patients will have baseline information collected and will complete baseline quality of life (QoL) questionnaires. QoL questionnaires will be obtained every 12 weeks +/- 2 weeks and survival will be measured through chart review. There will be no treatment intervention; however we will collect information on treatment received after enrolment in trial. Volume of leptomeningeal disease will be scored by number of gadolinium enhancing sites in 8 predetermined locations.

ELIGIBILITY:
Inclusion Criteria:

* Subject age is greater than or equal to 18 years at the time of signature of informed consent.
* Histologically or cytologically confirmed metastatic EGFR mutant NSCLC.
* Leptomeningeal disease based on brain MRI or CSF cytology.
* ECOG 0-3.
* Life expectancy of at least 8 weeks.
* Adequate hematologic and end organ function for testing.
* Ability to give informed consent for the study procedures defined in this protocol.

Exclusion Criteria:

* Inability to undergo a lumbar puncture due to thrombocytopenia, bleeding disorders, as well as inability to cooperate or consent to procedure.
* Subjects who are otherwise felt by the treating clinician to be unfit to proceed with this protocol.
* MRI spine demonstrating spinal leptomeningeal disease preventing a safe lumbar puncture.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2022-07-18 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Concordance of molecular profiling of CSF and plasma in EGFR mutation positive NSCLC patients with leptomeningeal disease | 36 months
  To determine the concordance rate of molecular alterations detected in the CSF and plasma of EGFR mutation positive NSCLC patients with leptomeningeal disease

SECONDARY OUTCOMES:
Concordance of treatment recommendations based on ctDNA and CSF | 36 months
  To determine the concordance and discordance between physician treatment recommendations based on ctDNA versus CSF molecular profiling.
Molecular profiling comparison | 36 months
  To assess concordance/discordance rates between ddPCR and Canexia Follow It completed on CSF and plasma based testing.
Molecular profiling descriptive comparison of patients treated with first/second generation versus 3rd generation EGFR TKIs | 36 months
  To identify molecular aberrations in the ctDNA and CSF of patients who progress on first/second EGFR TKIs and third generation EGFR TKIs to perform a descriptive comparison of shared and unique mutations identified based on prior exposure to first/second versus third generation EGFR TKI
Correlation between MRI and CSF | 36 months
  To correlate burden of leptomeningeal disease found on MRI and CSF positivity for tumor DNA.
Overall survival | 36 months
  To determine overall survival from time of developing leptomeningeal disease.
Quality of life with leptomeningeal disease | 36 months
  To assess the quality of life using the validated instrument, EuroQol 5 Dimension (EQ5D) (Scale of 0-100 where 0 is worst health and 100 is best health)

CONTACTS AND LOCATIONS:
Overall Officials: Cheryl Ho, MD, Principal Investigator — BC Cancer
Locations (1):
- BC Cancer, Vancouver, British Columbia, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Nevel KS, DiStefano N, Lin X, Skakodub A, Ogilvie SQ, Reiner AS, Pentsova E, Boire A. A retrospective, quantitative assessment of disease burden in patients with leptomeningeal metastases from non-small-cell lung cancer. Neuro Oncol. 2020 May 15;22(5):675-683. doi: 10.1093/neuonc/noz208. PMID 32352148
- [Background] White MD, Klein RH, Shaw B, Kim A, Subramanian M, Mora JL, Giobbie-Hurder A, Nagabhushan D, Jain A, Singh M, Kuter BM, Nayyar N, Bertalan MS, Stocking JH, Markson SC, Lastrapes M, Alvarez-Breckenridge C, Cahill DP, Gydush G, Rhoades J, Rotem D, Adalsteinsson VA, Mahar M, Kaplan A, Oh K, Sullivan RJ, Gerstner E, Carter SL, Brastianos PK. Detection of Leptomeningeal Disease Using Cell-Free DNA From Cerebrospinal Fluid. JAMA Netw Open. 2021 Aug 2;4(8):e2120040. doi: 10.1001/jamanetworkopen.2021.20040. PMID 34369989